CLINICAL TRIAL: NCT05173857
Title: Drug Eluting Balloon (DEB) vs Plain Old Balloon Angioplasty (POBA) for the Treatment of Failing Dialysis Access. A Prospective Randomized Trial
Brief Title: Drug Eluting Balloon (DEB) vs Plain Old Balloon Angioplasty (POBA) in the Treatment of Failing Dialysis Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Torbjorn Fransson, Consultant Vascular Surgeon, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TF1
Record Dates: First submitted 2021-11-10; First posted 2021-12-30 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Vascular Diseases; Kidney Diseases
Keywords: Haemodialysis; Fistula; Stenosis; Paclitaxel; Drug-eluting balloon; Angioplasty
MeSH Terms: conditions — Vascular Diseases; Kidney Diseases; Fistula; Constriction, Pathologic | interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Eluting Balloon (DEB) (Active Comparator): Percutaneous Angioplasty in dysfunctional arteriovenous access, using Drug Eluting Balloon Technology.
  Drug: Paclitaxel (PTX). Name of Device: Advance PTX
  Interventions: Device: Advance PTX; Drug: Paclitaxel (PTX)
- Plain Old Balloon Angioplasty (POBA) (Placebo Comparator): Percutaneous Angioplasty in dysfunctional arteriovenous access, using Plain Old Balloon Angioplasty.
  Drug: None. Name of Device: Advance LP (Low Profile)
  Interventions: Device: Advance LP (Low Profile)

INTERVENTIONS:
Device: Advance PTX — PTA in Dysfunctional Haemodialysis Access
  Arms: Drug Eluting Balloon (DEB)
Device: Advance LP (Low Profile) — Plain Old Balloon Angioplasty (POBA)
  Arms: Plain Old Balloon Angioplasty (POBA)
Drug: Paclitaxel (PTX) — Paclitaxel (PTX)
  Arms: Drug Eluting Balloon (DEB)

SUMMARY:
Background Conventional percutaneous transluminal angioplasty is still considered standard treatment for treatment of dysfunctional haemodialysis fistulas and grafts. The most important drawback with this treatment is frequent restenosis leading to a high number of secondary procedures. There is conflicting evidence in the literature regarding primary or secondary treatment with drug eluting balloons (DEB). These balloons deliver Paclitaxel locally, which acts as an antiproliferative drug and may improve treatment outcomes.

Methods This study was conducted as a prospective 1:1 randomized single centre clinical trial. Participants had primary or re-stenotic lesions in native upper extremity arteriovenous fistulas or at the graft-venous anastomosis. Patients were randomized to direct primary dilatation, with either a standard balloon or a DEB. The primary effectiveness endpoints were freedom from target lesion revascularization (TLR), access circuit revascularization or thrombosis, functional status of access circuit at 12 months. Secondary endpoints were procedural complications, procedural success, follow up survival and time to target lesion revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Active dialysis with a mature upper extremity dysfunctional haemodialysis access
* Primary stenosis or nonstented restenosis in a native AV fistula or at graft-venous location
* Adult (>18 years)
* Target vessel diameter 3-8mm

Exclusion Criteria:

* Thrombosed access
* In stent restenosis
* Pregnancy
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Freedom from restenosis in treated vascular access | 12 months
  Freedom from Restenosis and Target Lesion Revascularization (TLR) during 12 months follow up
Stenosis or occlusion in treated vascular access | 12 months
  Treated Denovo Stenosis or Occlusion during 12 months follow up, i.e a new stenosis >50%, not treated before in the study, and at another location in the vascular access circuit (upper arm haemodialysis access)
Number of Participants with a vascular access in full clinical use for haemodialysis at 12 months | 12 months
  Functional status of vascular access.